CLINICAL TRIAL: NCT06281743
Title: Attitudes to Decisions to Withdraw or Withhold Life-sustaining Treatments in Critically Ill Children- a Survey Among Pediatric Critical Care Physicians.
Brief Title: Attitudes to Decisions to Withdraw or Withhold Life-sustaining Treatments in Critically Ill Children
Acronym: LSTPedSurvey
Status: Active, not recruiting | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: LST-Ped Survey
Record Dates: First submitted 2024-01-16; First posted 2024-02-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Disorder; Critical Illness; Ethics, Narrative
MeSH Terms: conditions — Critical Illness; Narration | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — A web based survey is sent out to pediatric critical care physicians

SUMMARY:
The aim of this study is to investigate attitudes on decisions to withdraw or withhold life-sustaining treatments in critically ill children in Swedish intensive care units. This is a survey among pediatric critical care physicians.

DETAILED DESCRIPTION:
Sometimes, the best course of action for a patient is not to receive as much medical care as possible, but rather to prioritize other values. Making a decision to adjust the strategy and goals of care in this manner is referred to as a decision at the breaking point. A breaking point decision often involves decisions about treatment limitations. Treatment limitations in intensive care usually entail decisions to withhold or withdraw one or more life-sustaining treatments. Several events in Swedish society over the past decades may have influenced physicians' attitudes towards making decisions about withdrawing and withholding life-sustaining treatment. In 2009, a pediatric critical care physician was arrested for suspected manslaughter of a child in connection with the termination of intensive care. This initiated a protracted legal process in which the physician was acquitted but suffered significant personal harm due to false accusations. In 2011, the National Board of Health and Welfare issued updated regulations regarding life-sustaining treatments, followed by interpretations in guidelines and strategic documents in subsequent years. In 2020, the opportunity to donate organs was introduced not only after brain death diagnosis but also after circulatory arrest. The coronavirus infectious disease 2019 (COVID-19) pandemic emerged the same year. Sweden faced the threat of having to terminate intensive care not only for the patient's benefit but also due to resource constraints in intensive care. In 2019, a survey was conducted on end-of-life care decisions and practices from the perspective of personnel in pediatric intensive care in large parts of Europe. Sweden was not represented. The investigators are aware that Sweden stands out regarding socio-cultural values (http://www.worldvaluessurvey.org/). Since this has not been studied in Sweden before, and Sweden has a unique position regarding both traditional culture and an individual-centred societal view, it would be exciting to study the attitudes of physicians in Swedish intensive care units.

The investigators intend to map the attitudes of intensive care physicians regarding decisions to withhold/ and withdraw life-sustaining treatment in children within Swedish intensive care using an electronic survey. The method will be reported according to the checklist for reporting results of internet e-surveys (CHERRIES) checklist for web surveys. The survey will be explicitly designed for this study, incorporating a combination of new questions and questions previously used in similar surveys in other parts of Europe. The survey will be validated by a small group with expertise in the study subject and experience in survey research. Validity will be further confirmed through the calculation of Cronbach's alpha between the previously used questions and the new ones. Subsequently, a naive small test group will answer the survey and provide comments. Intensive care units with 10 or more instances of pediatric care visits lasting over 48 hours in 2023 will be selected. Data collection will occur by distributing a link to the web survey via email through a network of clinic managers at the selected intensive care units. It will be an open survey without control for duplicate responses and with a convenience sample. The survey introduction will provide information about the purpose of the study and how respondents' answers will be handled according to the General Data Protection Regulation (GDPR). Respondents will then confirm that they have understood the information before completing the survey. The response rate will be calculated as the proportion of completed surveys compared to the number of unique email addresses to which the survey link was sent. No checks for contradictory responses or incomplete surveys will be conducted before the respondent submits the survey. Incomplete surveys and surveys that take disproportionately long to complete will be analyzed. No propensity score matching or other weighting for differences will be performed. Data analysis will involve descriptive statistics, focusing on identifying correlations between respondents' attitudes toward withholding or withdrawing decisions, their clinical experiences, and any influential factors such as theoretical educational needs.

ELIGIBILITY:
Inclusion Criteria:

* Critical care physicians working with critically ill children in Swedish intensive care units

Exclusion Criteria:

* None

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Please
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Attitudes and experiences -questionnaire | 2024-2026
  Attitudes on decisions to withdraw or withhold life sustaining treatments in critically ill children in Swedish intensive care units. A questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Block, PhD, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: No